CLINICAL TRIAL: NCT03574012
Title: SmART Heart: Study of mHealth Apps to Reduce Cancer-Treatment Effects on the Heart
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 10037; NCI-2018-01168 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10037 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH); RG1001769 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2018-06-19; First posted 2018-06-29 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2020-09

CONDITIONS: Acute Leukemia in Remission; Hematopoietic Cell Transplantation Recipient; Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Monitoring, Physiologic

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (general health information, fitness tracker) (Active Comparator): Participants receive general information about physical activity and diet, and access to Fitbit and Healthwatch.
  Interventions: Device: Monitoring Device; Other: Informational Intervention; Other: Questionnaire Administration
- Intervention Group (individualized information, tracker) (Experimental): Participants receive individualized goal-setting and coaching in relation to physical activity and diet, supplemented with peer support through the study's social media platform, over 4 months. They also have access to mHealth apps including Fitbit and Healthwatch that provide feedback on physical activity and diet.
  Interventions: Device: Monitoring Device; Other: Informational Intervention; Other: Questionnaire Administration

INTERVENTIONS:
Device: Monitoring Device — Use Fitbit tracker
Other: Informational Intervention — Receive individualized health and fitness information from clinician, supplemented with peer support through the study's social media platform
  Arms: Intervention Group (individualized information, tracker)
Other: Informational Intervention — Receive general health and fitness information from clinician
  Arms: Control Group (general health information, fitness tracker)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This pilot trial studies how well education and mobile health applications work in reducing the effects of cancer treatment on the heart in participants with blood cancers that are in remission. Education and mobile health applications may be effective ways to manage heart health and to reduce future heart disease risk in participants with blood cancers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the feasibility of recruiting and retaining hematologic malignancy and hematopoietic cell transplantation (HCT) survivors in a randomized cardiovascular (CV) risk reduction mobile health (mHealth) counseling intervention.

II. Develop and refine a protocol to engage participants using an existing social medial platform and commercially available mHealth tools to reinforce lifestyle goals.

OUTLINE: Participants are randomized to 1 of 2 groups.

INTERVENTION GROUP: Participants receive individualized goal-setting and coaching in relation to physical activity and diet, supplemented with peer support through the study's social media platform, over 4 months. They also have access to mHealth apps including Fitbit and Healthwatch that provide feedback on physical activity and diet.

CONTROL GROUP: Participants receive general information about physical activity and diet, and access to Fitbit and Healthwatch.

After completion of study treatment, participants are followed up at 2 months and at 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Prior diagnosis of an acute leukemia or lymphoma or any receipt of HCT for a malignant condition.
* At time of approach, >= 5 years from initial cancer diagnosis or >= 5 years from first HCT, whichever is later.
* Currently in remission and not on any active anti-cancer therapies (survivors receiving maintenance tyrosine kinase inhibitors are NOT eligible).
* Able to read, write, and speak English.
* Access to smart phone or computer with internet access.
* Presence of at least 1 CV risk factor:

  * Currently on medication for hypertension, or
  * Currently on medication for cholesterol or triglyceride, or
  * Currently on medication for diabetes, or
  * Currently not physically active (self-reported average < 30 minutes/day), or
  * Currently smoking.
* Ability to understand and the willingness to provide informed consent.

Exclusion Criteria:

* Pre-existing ischemic heart disease (includes angina if documented in electronic medical record [EMR]) or ongoing symptomatic cardiomyopathy (those with asymptomatic cardiomyopathy may be allowed to participate if they do not have any current activity restrictions, but we will seek physician clearance for any submaximal exercise testing).
* Active systemic treatment for graft versus host disease.
* Currently pregnant. However, participants enrolled who become pregnant after randomization can remain on the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2018-08-31 (Actual); Primary Completion 2020-01-22 (Actual); Study Completion 2020-06-16 (Actual)

PRIMARY OUTCOMES:
Enrollment rate among participants approached | Up to 1 year
Retention rate among participants enrolled | Up to 1 year
  Retention is defined as completion of patient questionnaire and in-person assessment after 4-month intervention
Participation in Facebook group | Up to 1 year
  Number of participants who log onto the group page and participate at least one time (e.g., view a post, post something themselves, respond to a post [e.g., "like" a post], etc.)
Participation in Fitbit physical activity tracking | Up to 1 year
  Number of participants who submit step count data on at least 50% of eligible days
Participation in Healthwatch diet tracking | Up to 1 year
  Number of participants who provide dietary data on at least 75% of eligible days

CONTACTS AND LOCATIONS:
Overall Officials: Eric Chow, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

REFERENCES:
- [Result] Chow EJ, Doody DR, Di C, Armenian SH, Baker KS, Bricker JB, Gopal AK, Hagen AM, Ketterl TG, Lee SJ, Reding KW, Schenk JM, Syrjala KL, Taylor SA, Wang G, Neuhouser ML, Mendoza JA. Feasibility of a behavioral intervention using mobile health applications to reduce cardiovascular risk factors in cancer survivors: a pilot randomized controlled trial. J Cancer Surviv. 2021 Aug;15(4):554-563. doi: 10.1007/s11764-020-00949-w. Epub 2020 Oct 10. PMID 33037989